CLINICAL TRIAL: NCT01468363
Title: Hypervolemia and Treatment Guided by Bioimpedance in End Stage Renal Disease Patients in Zonguldak (Prospective Study)
Brief Title: Hypervolemia in ESRD Patients in Zonguldak (Prospective Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Ender Hur, Medical Doctor, Specialist, Nephrology Department, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKU 2011-77-21/06
Record Dates: First submitted 2011-11-05; First posted 2011-11-09 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Hemodialysis Fluid Allergy
Keywords: Dry weight; Body composition monitor; Hemodialysis; Zonguldak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): "Overhydration (OH) in liters" will be estimated with the BCM (Body Composition Monitor, Fresenius Medical Care, Deutschland GmbH) in order to determine dry weight as needed before a dialysis session.
  1. If OH is positive value, we will try to reach dry weight by ultrafiltration without regard to the level of blood pressure.
  2. If OH is negative value , we will not change dry weight.
  Interventions: Device: Dry weight adjustment
- Group 2 (No Intervention): BCM results obtained at the beginning and 12th months will not be given to the treating physicians. Dry weight estimation will be guided by clinical findings, telecardiography, and echocardiography as used to be.
  Interventions: Device: Dry weight adjustment

INTERVENTIONS:
Device: Dry weight adjustment — Dry weight adjustment according to BCM results
  Other Names: Group 1: BCM Adjusted Group; Group 2: Classical Group

SUMMARY:
There is no easily applicable method to determine extra cellular volume and consequently estimate DW. Thus DW has to be clinically defined by ''trial and error'' and several indirect methods.

Recently, devices to measure DW by Bioimpedance spectroscopy (BİS) have become available. This non-invasive, cheap easily repeatable method has the potential to improve dialysis outcome in the majority of patients all over the world, The aim of the present project is to assess the feasibility of volume control by using a BİS device.

DETAILED DESCRIPTION:
The excessive mortality of dialysis patients, particularly from cardiovascular events, is undoubtedly related for a large part to hypertension and cardiac damage(1). Most studies reveal that hypertension persists despite antihypertensive drugs. Some authors (Parfrey) have used the term ''natural history'' of heart disease in dialysis, suggesting that deterioration is inevitably linked to that procedure (2).

In sharp contrast, other studies (Charra, Özkahya)(3,4) have shown that a strict volume control strategy decreases blood pressure (BP) without drugs, and prolongs survival. This suggests that volume control is insufficient in most dialysis centers, despite the fact that treating physicians may consider that ''Dry Weight'' (DW) of their patients has been reached. In fact, there is no easily applicable method to determine extra cellular volume and consequently estimate DW. Thus DW has to be clinically defined by ''trial and error'' and several indirect methods.

Recently, devices to measure DW by Bioimpedance spectroscopy (BİS) have become available. This non-invasive, cheap easily repeatable method has the potential to improve dialysis outcome in the majority of patients all over the world, The aim of the present project is to assess the feasibility of volume control by using a BİS device and compare the results with the conventional ways of treatment.

Conventional ways to estimate DW (5)Intradialytic hypotension continues to be a leading problem, especially in the elderly and cardiovascularly compromised patient. This predominance can be explained by the fact that structural and functional abnormalities of the heart and blood vessels increase the sensitivity of the patient to changes in fluid status. It does not only cause discomfort, but also increases mortality. In a recent study, a low post-dialytic blood pressure was associated with a significantly increased risk for mortality . Therefore prevention of intradialytic hypotension, remains an important challenge to the dialysis physician.

The occurrence of hypotension during ultrafiltration (UF) necessitates termination of the UF procedure and is commonly considered as a sign that DW has been reached. However, although intradialytic hypotension is commonly considered to be a sign of hypovolemia, this is not always correct, because too rapid removal of large amounts of fluid within a few hours causes a temporary state of disequilibrium. It has been shown that achievement of DW by volume control in fact decreases the number of hypotensive episodes (5) Therefore, there is a need for objective methods to estimate the body fluid volumesThis prospective, randomized, controlled study aims to evaluate the usefulness of the new BCM device as a method to improve volume control dialysis patients and compare the results with those obtained by conventional volume control modalities. To our knowledge such an investigation has not been done elsewhere.

The investigators believe that the proposed study will produce powerful evidence to convince the nephrological society of the need for strict volume control strategy by using new device BCM in hemodialysis patients. The expected data may change routine practice causing achievement of normal blood pressure level without using anti-hypertensive medication.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18-year,
* Maintenance bicarbonate HD scheduled thrice weekly (12 hours/week),
* Willingness to participate in the study with a written informed consent.

Exclusion Criteria:

* Presence of a cardiac stent, pacemaker or defibrillator ,
* Artificial joints, pin or amputation
* Permanent or temporary catheters (may affect BCM measurement),
* Beeing scheduled for living donor renal transplantation,
* Presence of serious life-limiting co-morbid situations, like malignancy, uncontrollable infection, end-stage cardiac, pulmonary, or hepatic disease,
* Pregnancy or lactating,
* Current use of investigational drugs or participation in an interventional clinical trial that contradicts or interferes with the therapies or measured outcomes in this trial,
* Mental incompetence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Evidence of hypervolemia confirmed by non-invasive bioimpedance spectroscopy technique | within 1 year

SECONDARY OUTCOMES:
Achievement of normal blood pressure level without using anti-hypertensive medication | within 1 year
  Achievement of normal blood pressure level without using anti-hypertensive medication Changes in post-dialysis body weight Hematocrit and related rHu-EPO doses Serum levels of albumin and Hs-CRP

CONTACTS AND LOCATIONS:
Overall Officials: Ender Hur, M.D, Principal Investigator — ZKU Nephrology Department
Locations (10):
- Turkey (Türkiye) (10):
  - Devrek Devlet Hastanesi, Zonguldak, Devrek
  - Ereğli Devlet Hastanesi Diyaliz Merkezi, Zonguldak, Ereğli
  - Ereğlı Burcu Koç Diyaliz Merkezi, Zonguldak, Ereğli
  - Ereğlı Can Diyaliz Merkezi, Zonguldak, Ereğli
  - Atatürk Devlet Hastanesi Diyaliz Merkezi, Zonguldak
  - Devrek Can Diyaliz Merkezi, Zonguldak
  - ZKU Uygulama ve Arş Hastanesi Diyaliz Merkezi, Zonguldak
  - Zonguldak Can Diyaliz Merkezi, Zonguldak
  - Çaycuma Devlet Hastanesi Diyaliz Merkezi, Zonguldak
  - Çaycuma Can Diyaliz Merkezi, Zonguldak, Çaycuma

REFERENCES:
- [Result] Akcicek F, Dilber S, Ozgen G, Ok E, Akalin E, Atabay G, Basci A, Guclu A, Dorhout Mees EJ. Spontaneous perirenal hematoma due to periarteritis nodosa. Nephron. 1994;68(3):396. doi: 10.1159/000188413. No abstract available. PMID 7838273
- [Result] Coker A, Ok E, Tokat Y, Hoscoskun C, Kaplan H, Yararbas O. Evaluation of patients transplanted in countries other than Turkey. Transplant Proc. 1994 Aug;26(4):2455-6. No abstract available. PMID 8066803
- [Result] Ok E, Akcicek F, Toz H, Kursat S, Tobu M, Basci A, Mees EJ. Comparison of the effects of enalapril and theophylline on polycythemia after renal transplantation. Transplantation. 1995 Jun 15;59(11):1623-6. PMID 7778179
- [Result] Ok E, Akcicek F, Coker A, Tombuloglu M, Toz H, Tokat Y, Cirit M, Tobu M, Onder G, Basci A. Alloimmune haemolytic anaemia after renal transplantation. Nephrol Dial Transplant. 1995;10(3):404-5. No abstract available. PMID 7792041
- [Result] Ok E, Akcicek F, Dorhout Mees EJ, Basci A, Mir S, Kursat S, Unsal A. Malignant hypertension in a haemodialysis patient treated by ultrafiltration. Nephrol Dial Transplant. 1995 Nov;10(11):2124-5. No abstract available. PMID 8643182